CLINICAL TRIAL: NCT01431664
Title: A Cancer Research UK Phase I/IIa Trial of AT9283 (A Selective Inhibitor of Aurora Kinases) Given Over 72 Hours Every 21 Days Via Intravenous Infusion in Children and Adolescents Aged 6 Months to 18 Years With Relapsed and Refractory Acute Leukemia
Brief Title: AT9283 in Treating Young Patients With Relapsed or Refractory Acute Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000709775; CRUK-CR0708-12; EUDRACT-2009-016952-36
Record Dates: First submitted 2011-09-08; First posted 2011-09-09 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; acute leukemias of ambiguous lineage; acute undifferentiated leukemia; secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute

INTERVENTIONS:
Drug: multikinase inhibitor AT9283
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: AT9283 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I/IIa clinical trial is studying the side effects and best dose of AT9283 in treating young patients with relapsed or refractory acute leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To identify the maximum-tolerated dose and recommended phase IIb dose of multikinase inhibitor AT9283 in pediatric patients with relapsed or refractory acute leukemia.

Secondary

* To evaluate the safety and tolerability of this drug in these patients.
* To document evidence of efficacy of this drug in these patients.
* To investigate the pharmacokinetic profile of this drug in plasma in these patients.

Tertiary

* To assess target kinase inhibition by multikinase inhibitor AT9283 in these patients.
* To identify potential predictive molecular biomarkers in these patients.

OUTLINE: This is a multicenter study.

Patients receive multikinase inhibitor AT9283 IV continuously over 72 hours. Treatment repeats every 21 days* for 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving benefit of treatment may continue for up to 6 more courses at the discretion of the chief/principal investigator.

NOTE: *Course length may be extended to a maximum 42 days to allow for recovery of blood counts. Intrathecal therapy is permitted from course 2 onwards in patients with ALL.

Blood specimens are collected for pharmacokinetic and pharmacodynamic studies including molecular predictive biomarkers and ex vivo and in vivo measurement of kinase inhibition assessments.

After completion of study treatment, patients are followed up for 42 days or until recovery of blood counts (whichever is the sooner).

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute leukemia according to the following criteria:

  * Acute lymphoblastic leukemia (ALL) meeting any of the following criteria:

    * Second relapse
    * Refractory to induction therapy for first relapse
    * Third or subsequent relapse
  * Acute myeloid leukemia (AML) meeting any of the following criteria:

    * Second or subsequent relapse
    * Refractory to an induction therapy for first relapse
    * Without a curative treatment option
  * Other type of acute leukemia meeting any of the following criteria:

    * First or subsequent relapse
    * Refractory to induction therapy
    * Not eligible for any therapy of higher curative potential
* No chronic myeloid leukemia (CML)
* Patients in relapse must have ≥ 5% blasts in the bone marrow
* Patients with refractory disease following induction must have ≥ 20% blasts in the bone marrow
* No evidence of CNS disease

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% OR Lansky PS 50-100%
* Life expectancy ≥ 8 weeks
* Serum bilirubin < 1.5 times upper limit of normal (ULN)
* ALT or AST < 2.5 times ULN (5 times ULN if due to leukemic infiltration of the liver)
* Creatinine clearance ≥ 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use 2 of the following combined forms of contraception (oral, injected, or implanted hormonal contraception and condom OR intra-uterine device and condom OR diaphragm with spermicidal gel and condom) before, during, and for 6 months after completion of study therapy
* Male patients must use 1 form of highly effective contraception (condom plus spermicidal gel) during and for 6 months after completion of study therapy

  * Men with pregnant or lactating partners should be advised to use barrier-method contraception (condom plus spermicidal gel)
* No serological positivity for hepatitis B, hepatitis C, or HIV
* No congenital heart disease, with the exception of patent foramen ovale or small muscular ventricular septal deficit (within the first year of life)
* No uncontrolled arterial hypertension (defined as a systolic blood pressure [BP] and/or diastolic BP ≥ 95th percentile for age and height)
* No fractional shortening of ≤ 29% on echocardiogram
* No active graft-vs-host disease
* No current non-malignant systemic disease considered high medical risk, including any of the following:

  * Active uncontrolled infection
  * Unstable or uncompensated respiratory or cardiac condition that makes study participation undesirable
* No other condition that, in the Investigator's opinion, would not make the patient a good candidate for the clinical trial

PRIOR CONCURRENT THERAPY:

* Recovered from toxicity of prior therapy, including toxicity following hematopoietic stem cell transplantation

  * Alopecia or certain grade 1 toxicities allowed at the discretion of the Investigator
* A maximum of 2 days of hydroxycarbamide 10-20 mg/kg/day (or according to local practice) in patients with AML and hyperleukocytosis allowed
* At least 7 days since prior investigational drugs (except antibodies for which a 4-week window must be observed)
* At least 7 days since prior protein kinase inhibitors and intrathecal therapy

  * Concurrent intrathecal therapy allowed from course 2 onwards in patients with ALL
* At least 14 days since prior cytotoxic therapy, including vincristine and other anti-neoplastics
* No prior major thoracic or abdominal surgery from which the patient has not yet recovered
* No prior aurora kinase inhibitor
* No concurrent steroid therapy

  * Multikinase inhibitor AT9283 administration may be commenced once steroids have started; however, steroids may not be started once multikinase inhibitor AT9283 has started
  * Up to 5 days of prior oral dexamethasone (6 mg/m^2) for patients with ALL experiencing a rapid rise in blast count allowed
* No other concurrent interventional clinical study

  * Participation in an observational study allowed
* No other concurrent anticancer therapy or investigational drugs

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2011-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose and recommended phase II dose of multikinase inhibitor AT9283

SECONDARY OUTCOMES:
Adverse events to multikinase inhibitor AT9283 and grading severity according to NCI CTCAE Version 4.02
Partial remission, complete remission, or complete remission with incomplete bone marrow recovery using disease-specific criteria based on ANC, platelets, and % blasts in the bone marrow
Plasma concentration measurement of multikinase inhibitor AT9283
Tertiary outcome(s) - Ex vivo and in vivo measurement of kinase inhibition using Plasma Inhibitory Activity (PIA) assay, phosphorylated STAT5 assay, and skin-punch biopsy (measuring pHH3, p53, PCNA, Ki67 levels)
Results of established and novel prognostic biomarkers (genetic mutations of JAK 1, 2, 3, FLT3, IKAROS, and BCR/ABL) linking to observed responses

CONTACTS AND LOCATIONS:
Overall Officials: Josef Vormoor, Principal Investigator — Sir James Spence Institute of Child Health at Royal Victoria Infirmary
Locations (5):
- United Kingdom (5):
  - Royal Marsden Hospital, Surrey, London
  - Birmingham Children's Hospital, Birmingham
  - Leeds General Infirmary, Leeds
  - Royal Manchester Children's Hospital, Manchester
  - Great North Children's Hospital, Royal Victoria Infirmary, Newcastle upon Tyne